CLINICAL TRIAL: NCT01337726
Title: Combined Illness Management and Psychotherapy in Treating Depressed Elders
Acronym: COPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn L Turvey, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH086482 (NIH); R01MH086482 (NIH)
Record Dates: First submitted 2011-03-24; First posted 2011-04-19 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2016-05

CONDITIONS: Depression; Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Depression; Heart Failure; Chronic Obstructive Pulmonary Disease; Quality of Life; Functional Impairment
MeSH Terms: conditions — Depression; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Illness Management Only (Active Comparator)
  Interventions: Behavioral: Illness Management Only
- Combined Psychotherapy & Illness Management (Experimental)
  Interventions: Behavioral: Combined Psychotherapy and Illness Management

INTERVENTIONS:
Behavioral: Combined Psychotherapy and Illness Management — Participants will have 10 weekly visits with a study clinician at their home and by phone. They will focus on their self care and illness management as well as how to manage their mood/cope emotionally. Follow up assessments will occur at 26 and 52 weeks.
  Arms: Combined Psychotherapy & Illness Management
Behavioral: Illness Management Only — Participants in this group will have 10 weekly sessions with a study clinician at home and by phone. They will focus only on how they manage their illness. Follow up assessments will occur at 26 and 52 weeks.
  Arms: Illness Management Only

SUMMARY:
The purpose of this research study is to test a program developed to help patients with chronic heart or lung problems take care of themselves and cope with their illness or limitations.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years or older
* Diagnosis of Heart Failure or COPD
* Depressive symptoms indicated by a BDI-II score of 10 or higher
* Functional impairment

Exclusion Criteria:

* Current psychotherapy
* Cognitive Impairment
* Psychiatric diagnosis
* Active suicidal thoughts
* Significant vision or hearing impairment
* Residence in long term care facility

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2011-02; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | 10 weeks
  Change from Baseline in depressive symtoms at 10 weeks

SECONDARY OUTCOMES:
Improvement in quality of life/functioning | 10 weeks
  Change from Baseline in quality of life/functioning at 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn L. Turvey, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - Iowa City VA Health Care System, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa